CLINICAL TRIAL: NCT02481375
Title: Is Iron Deficiency the Cause of Anemia Among Women of Reproductive Age in Cambodia? A 2 x 2 Factorial Double Blind Randomized Controlled Trial of Oral Iron and Multiple Micronutrient Supplementation
Brief Title: Is Iron Deficiency the Cause of Anemia Among Women in Cambodia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Micronutrient Initiative (Other); DSM Nutritional Products, Inc. (Industry); International Development Research Centre, Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); Helen Keller International (Other)
Responsible Party: Principal Investigator, Tim Green, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: H15-00933
Record Dates: First submitted 2015-06-10; First posted 2015-06-25 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Anemia; Iron Deficiency; Hemoglobin Disorder; Infection; Inflammation
Keywords: iron; ferritin; soluble transferrin receptor; hepcidin; reticulocyte count; hemoglobin; supplementation
MeSH Terms: conditions — Anemia; Iron Deficiencies; Hemoglobinopathies; Infections; Inflammation | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Multiple micronutrients with iron (Experimental): Multiple micronutrient formulations were based on the UNICEF/WHO/UNU standard formulation for pregnant and lactating women (UNIMMAP) with increased iron (from 30 mg to 60 mg elemental iron) for comparability to the iron only group (60 mg). This formulation has 15 micronutrients including iron.
  Women will receive the multiple micronutrient with iron for 12 weeks.
  Interventions: Dietary Supplement: Multiple micronutrients; Dietary Supplement: Iron
- Multiple micronutrients without iron (Active Comparator): This formulation has the 14 micronutrients included in the UNIMMAP formulation, but does not include iron.
  Women will receive the multiple micronutrient without iron for 12 weeks.
  Interventions: Dietary Supplement: Multiple micronutrients
- Iron only (Active Comparator): This formulation only has 60 mg elemental iron.
  Women will receive iron for 12 weeks.
  Interventions: Dietary Supplement: Iron
- Placebo (Placebo Comparator): This formulation is a placebo.
  Women will receive a placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multiple micronutrients — 12-wk supplementation of vitamin A, B1, B2, B6 ,B12, D, E, niacin, folic acid, zinc, copper, selenium, iodine
  Arms: Multiple micronutrients with iron; Multiple micronutrients without iron
Dietary Supplement: Iron — 12-wk supplementation of iron
  Other Names: 60 mg elemental iron
  Arms: Iron only; Multiple micronutrients with iron
Dietary Supplement: Placebo — 12-wk supplementation of placebo
  Arms: Placebo

SUMMARY:
Globally, the most common cause of anemia is thought to be iron deficiency anemia (IDA). This was assumed to be the major cause of anemia in Cambodia, because Cambodian diets, which consist mainly of rice, lack iron-rich animal food sources. However, our findings from a previous study in Cambodia (a Canadian government funded study investigating multiple interventions to improve food and nutrition security) showed that IDA is almost non-existent and challenges this assumption. In a cross-sectional survey of 450 women from rural Cambodia, only 1.0% had Hb and ferritin levels indicative of IDA (Hb <120 g/L and ferritin <15 μg/L). A national survey conducted by UNICEF in 2014 found similarly low rates of IDA (Dr. Arnaud Laillou, UNICEF Cambodia). Further, other micronutrients known to be associated with anemia were also low (<3%) including folate and vitamins B12 and B6.

In addition, 54% of the Prey Veng women had a genetic Hb disorder (e.g., α-thalassemias), which are inherited diseases that can result in a defective Hb structure and/or impair Hb production, either of which can reduce Hb concentration and increase the risk of anemia. Further, genetic Hb disorders cause ferritin and soluble transferrin receptor (sTfR) concentrations to increase, which reduce the diagnostic sensitivity of these biomarkers to identify IDA.

In 2011, the Cambodian Ministry of Health (MOH) recommended weekly iron and folic acid (IFA) supplementation for all women of reproductive age, consistent with WHO guidelines. However, if iron deficiency is not a major cause of anemia, then at best supplementation is a waste of valuable resources and at worst could cause harm. Further, the justification for provision of multiple micronutrients among this population has not yet been proven, despite the push from some organizations such as the WHO. There is an urgent need to conduct a trial to clarify whether iron or other micronutrient deficiencies are a major cause of anemia in Cambodia.

Research Objectives:

1. To compare Hb concentration (g/L) after 12-weeks of supplementation in women to determine if iron significantly improves Hb concentration, compared to a placebo;
2. To compare Hb concentration (g/L) across the four groups (multiple micronutrients with iron, multiple micronutrients without iron, iron alone, and placebo) after 12-weeks; and
3. To determine which of the hematological indicators (ferritin, sTfR, reticulocyte count and hepcidin) have the strongest diagnostic ability to predict responsiveness to iron therapy after 12-weeks using receiver operating characteristic (ROC) analyses.

Methods: A 2 x 2 factorial randomized controlled trial will be conducted over 12 weeks. A total of ~800 women (18-45 y) with mild or moderate anemia will be recruited and randomized to 1 of 4 groups: multiple micronutrients with iron, multiple micronutrients without iron, iron alone or placebo. Blood will be collected at baseline and at 1 and 12 weeks after the intervention and assessed for Hb, hematological biomarkers, inflammation and genetic Hb disorders. The investigators will use a general linear model to measure differences in Hb concentration across the four groups after the intervention. Receiver operating characteristic curves will be used to determine the diagnostic ability of the multiple hematological indicators to predict responsiveness to iron therapy.

DETAILED DESCRIPTION:
Background:

Anemia is a severe public health problem in Cambodia, affecting ~44% of women of reproductive age. Defined as a hemoglobin (Hb) concentration below 120 g/L, anemia can increase the risk of adverse pregnancy outcomes and impair work capacity and productivity. The potential causes of anemia are poor nutrition (e.g. micronutrient deficiencies), genetic Hb disorders (e.g. thalassemia), and inflammation and disease.

Globally, the most common cause of anemia is thought to be iron deficiency anemia (IDA). This was assumed to be the major cause of anemia in Cambodia, because Cambodian diets, which consist mainly of rice, lack iron-rich animal food sources. However, our findings from a previous study in Cambodia (a Canadian government funded study investigating multiple interventions to improve food and nutrition security) showed that IDA is almost non-existent and challenges this assumption. In a cross-sectional survey of 450 women from rural Cambodia, only 1.0% had Hb and ferritin levels indicative of IDA (Hb <120 g/L and ferritin <15 μg/L). A national survey conducted by UNICEF in 2014 found similarly low rates of IDA (Dr. Arnaud Laillou, UNICEF Cambodia). Further, other micronutrients known to be associated with anemia were also low (<3%) including folate and vitamins B12 and B6. On the other hand, other nutrients known to be associated with anemia such as zinc and riboflavin deficiencies were prevalent (30% and 82%, respectively). In addition, 54% of the Prey Veng women had a genetic Hb disorder (e.g., α-thalassemias), which are inherited diseases that can result in a defective Hb structure and/or impair Hb production, either of which can reduce Hb concentration and increase the risk of anemia. Further, genetic Hb disorders cause ferritin and soluble transferrin receptor (sTfR) concentrations to increase, which reduce the diagnostic sensitivity of these biomarkers to identify IDA.

In 2011, the Cambodian Ministry of Health (MOH) recommended weekly iron and folic acid (IFA) supplementation for all women of reproductive age, consistent with WHO guidelines. However, if iron deficiency is not a major cause of anemia, then at best supplementation is a waste of valuable resources and at worst could cause harm. Further, the justification for provision of multiple micronutrients among this population has not yet been proven, despite the push from some organizations such as the WHO. There is an urgent need to conduct a trial to clarify whether iron or other micronutrient deficiencies are a major cause of anemia in Cambodia.

Research Hypotheses:

The iron-supplemented group will have a significantly higher mean Hb concentration than the placebo group after 12-weeks, indicating a higher prevalence of iron deficiency than suggested by ferritin and sTfR biomarkers at baseline. The multiple micronutrients with iron group will have a significantly higher mean Hb concentration than the iron alone-supplemented group, indicating that the addition of other micronutrients confer a benefit in reducing anemia. Reticulocyte count is the most sensitive biomarker to predict the responsiveness to iron therapy.

Research Goals and Objectives:

Goal 1. To determine if iron deficiency exists among women in Cambodia, where genetic Hb disorders and inflammation are prevalent, by conducting a randomized controlled trial of iron supplementation.

Objective 1: To compare Hb concentration (g/L) after 12-weeks of supplementation in women to determine if iron significantly improves Hb concentration, compared to a placebo.

Goal 2: To determine if the addition of other micronutrients confers any additional benefit to iron supplementation, by conducting a 2 x 2 factorial study design.

Objective 2: To compare Hb concentration (g/L) across the four groups (multiple micronutrients with iron, multiple micronutrients without iron, iron alone, and placebo) after 12-weeks.

Goal 3. To investigate multiple biomarkers of iron deficiency to determine which is most sensitive and specific to predict the response to iron or multiple micronutrient with iron supplementation.

Objective 3: To determine which of the hematological indicators (baseline values for ferritin, sTfR, reticulocyte count and hepcidin) have the strongest diagnostic ability to predict responsiveness to iron therapy after 12-weeks using receiver operating characteristic (ROC) analyses.

Study Design:

A 2 x 2 factorial double blind randomized controlled trial will be conducted over 12 weeks. A total of ~800 women (18-45 y) with anemia will be recruited and randomized to 1 of 4 groups: multiple micronutrients with iron, multiple micronutrients without iron, iron alone or placebo.

Population and Setting: Cambodian women will be recruited to local health centers using convenience sampling from 4 randomly selected villages in a peri-urban area of Kampong Chhnang province. This province is ~1.5 hours outside of the capital city of Phnom Penh.

Randomization: Women will be randomized 1:1 by a computer-generated random list to one of four interventions (n=200 each group). Randomization to either a treatment or control group will reduce bias and confounding factors, which may affect the Hb response (outcome). The manufacturers of the gel capsules will be responsible for blinding the four interventions at time of capsule packaging and will retain confidentiality of capsule contents until the time of study completion.

Methods:

Blood will be collected at baseline, and at 1 and 12 weeks after the intervention and assessed for Hb, hematological biomarkers (reticulocyte count, MCV, RDW, hepcidin), micronutrients and iron biomarkers (vitamin B12, folate, zinc, riboflavin, ferritin, sTfR, RBP) inflammation (AGP and CRP) and genetic Hb disorders. We will use a general linear model to measure differences in Hb concentration across the four groups after the intervention. Receiver operating characteristic curves will be used to determine the diagnostic ability of the multiple hematological indicators to predict responsiveness to iron therapy.

Implications: This translational research is urgently required in Cambodia to build the evidence needed to inform the Ministry of Health on strategies, policy and programs to reduce, prevent and treat anemia among women in Southeast Asia (~300,000,000) and among Southeast Asian immigrants in Canada (who will number ~450,000 by 2031).

ELIGIBILITY:
Inclusion Criteria:

1. women between 18-45 years
2. healthy except for Hb = or <117 g/L
3. consent to participate in the study.

Exclusion Criteria:

1. women with Hb >117 g/L
2. women who are currently pregnant
3. women who are taking medications, including any dietary supplements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 809 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kroeun Hou, MPH, Study Chair — Helen Keller International, Cambodia; Sophonneary Prak, MPH, Study Chair — National Maternal and Child Health Center, Ministry of Health, Cambodia; Crystal Karakochuk, MSc, PhD(c), Study Chair — University of British Columbia; Tim Green, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Kampong Chhnang province, Kampong Chhnang, Kampong Chhnang, Cambodia

REFERENCES:
- [Derived] Williams BA, Cochrane KM, Fischer JAJ, Aljaadi AM, McAnena L, Ward M, McNulty H, Kroeun H, Green TJ, Whitfield KC, Karakochuk CD. The Homozygous Hemoglobin EE Variant Is Associated with Poorer Riboflavin Status in Cambodian Women of Reproductive Age. J Nutr. 2020 Jul 1;150(7):1943-1950. doi: 10.1093/jn/nxaa119. PMID 32433728
- [Derived] Holmes JB, Kroeun H, Houghton LA, Gibson RS, Harding KB, De-Regil LM, Kraemer K, Barr SI, Karakochuk CD. Including 60 mg Elemental Iron in a Multiple Micronutrient Supplement Blunts the Increase in Serum Zinc after 12 Weeks of Daily Supplementation in Predominantly Anemic, Nonpregnant Cambodian Women of Reproductive Age. J Nutr. 2019 Sep 1;149(9):1503-1510. doi: 10.1093/jn/nxz097. PMID 31174215
- [Derived] Karakochuk CD, Barker MK, Whitfield KC, Barr SI, Vercauteren SM, Devlin AM, Hutcheon JA, Houghton LA, Prak S, Hou K, Chai TL, Stormer A, Ly S, Devenish R, Oberkanins C, Puhringer H, Harding KB, De-Regil LM, Kraemer K, Green TJ. The effect of oral iron with or without multiple micronutrients on hemoglobin concentration and hemoglobin response among nonpregnant Cambodian women of reproductive age: a 2 x 2 factorial, double-blind, randomized controlled supplementation trial. Am J Clin Nutr. 2017 Jul;106(1):233-244. doi: 10.3945/ajcn.116.140996. Epub 2017 May 10. PMID 28490515
- [Derived] Rappaport AI, Barr SI, Green TJ, Karakochuk CD. Variation in haemoglobin measurement across different HemoCue devices and device operators in rural Cambodia. J Clin Pathol. 2017 Jul;70(7):615-618. doi: 10.1136/jclinpath-2017-204351. Epub 2017 Mar 8. PMID 28275044

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Micronutrients With Iron: Multiple micronutrient formulations were based on the UNICEF/WHO/UNU standard formulation for pregnant and lactating women (UNIMMAP) with increased iron (from 30 mg to 60 mg elemental iron) for comparability to the iron only group (60 mg). This formulation has 15 micronutrients including iron.
  Women will receive the multiple micronutrient with iron for 12 weeks.
  Multiple micronutrients: 12-wk supplementation of vitamin A, B1, B2, B6 ,B12, D, E, niacin, folic acid, zinc, copper, selenium, iodine
  Iron: 12-wk supplementation of iron
- Multiple Micronutrients Without Iron: This formulation has the 14 micronutrients included in the UNIMMAP formulation, but does not include iron.
  Women will receive the multiple micronutrient without iron for 12 weeks.
  Multiple micronutrients: 12-wk supplementation of vitamin A, B1, B2, B6 ,B12, D, E, niacin, folic acid, zinc, copper, selenium, iodine
- Iron Only: This formulation only has 60 mg elemental iron.
  Women will receive iron for 12 weeks.
  Iron: 12-wk supplementation of iron
- Placebo: This formulation is a placebo.
  Women will receive a placebo for 12 weeks.
  Placebo: 12-wk supplementation of placebo
Period: Overall Study
Arm/Group | Multiple Micronutrients With Iron | Multiple Micronutrients Without Iron | Iron Only | Placebo
Started | 206 | 202 | 201 | 200
Completed | 192 | 191 | 191 | 186
Not Completed | 14 | 11 | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple Micronutrients With Iron | Multiple Micronutrients Without Iron | Iron Only | Placebo | Total
Number analyzed (Participants) | 206 | 202 | 201 | 200 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] — Verified that the Standard Deviation values were identical for all Arms/Groups.
  years | 30 (8) | 30 (8) | 31 (8) | 30 (8) | 30 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 202 | 201 | 200 | 809
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Cambodia | 206 | 202 | 201 | 200 | 809

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Levels at 12-weeks. Marginal Means (95% CI).
Description: Marginal means (95% CI) at 12-weeks using a generalized mixed-effects model with adjustments for baseline values and village clusters. Multiple imputation was used to impute n=49 missing values for hemoglobin at endline.
Time Frame: 12-weeks of intervention
Measure: Mean (95% Confidence Interval); unit: g/L
Arm/Group | Multiple Micronutrients With Iron | Multiple Micronutrients Without Iron | Iron Only | Placebo
Number analyzed (Participants) | 206 | 202 | 201 | 200
g/L | 123 [122 to 123] | 116 [116 to 117] | 121 [120 to 121] | 116 [116 to 117]
Statistical Analysis 1: Comparison: Multiple Micronutrients With Iron vs Multiple Micronutrients Without Iron vs Iron Only vs Placebo; Marginal means (95% CI) of ferritin concentrations at 12-weeks using a generalized mixed-effects model with adjustments for baseline values and village clusters; Test type: Other; p < 0.05, Regression, Linear; Marginal means = 0

ADVERSE EVENTS:
Time Frame: 12-weeks
Description: Adverse events were reported as combined (any of the following) - GI distress, constipation, vomiting, and diarrhea.
Arm/Group | Multiple Micronutrients With Iron | Multiple Micronutrients Without Iron | Iron Only | Placebo
Serious Adverse Events (participants affected / at risk) | 138/200 | 103/195 | 101/197 | 86/197
Other Adverse Events (participants affected / at risk) | 0/200 | 0/195 | 0/197 | 0/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Micronutrients With Iron (N=200) | Multiple Micronutrients Without Iron (N=195) | Iron Only (N=197) | Placebo (N=197)
Adverse side effects (GI distress, constipation, vomiting, diarrhea) (Gastrointestinal disorders) | 138 (138) | 103 (103) | 101 (101) | 86 (86)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No